CLINICAL TRIAL: NCT05379244
Title: Better Sleep in Psychiatric Care - Clinical Feasibility and Preliminary Effects of CBT for Insomnia in a Mixed Psychiatric Sample at an Outpatient Clinic
Brief Title: Better Sleep in Psychiatric Care - Depression, Anxiety and Trauma, Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Susanna Jernelöv, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/80-31/1a
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Anxiety Disorders; Affective Disorders; PTSD; Insomnia Chronic
Keywords: CBT-i
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Pragmatic, within-group pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT-i (Experimental): Cognitive Behavioral Therapy for insomnia adjusted for patients with mixed psychiatric disorders
  Interventions: Behavioral: CBT-i

INTERVENTIONS:
Behavioral: CBT-i — Behavioral intervention based on Cognitive Behavioral Therapy for insomnia, adjusted for psychiatric patients with anxiety disorders, affective disorders and trauma

SUMMARY:
Between 50-80 percent of patients in psychiatry have insomnia-type sleep problems. In addition to reduced quality of life and impaired function, sleep problems can aggravate other psychiatric problems and increase the risk of relapse into, for example, depression. According to international guidelines, cognitive behavioral therapy for insomnia (CBT-i) should be used as the first choice for treatment of insomnia. In practice, however, it is very uncommon for psychiatric patients to be offered CBT-i, instead most are treated with sleep medications. There is also a lack of research studies evaluating CBT-i in regular clinical practice.

This pilot study investigated the feasibility of a group treatment with CBT-i at a psychiatric outpatient clinic in Stockholm for patients with depression, bipolar disorder II, anxiety syndrome and PTSD. Changes in symptoms of insomnia, depression, and anxiety after treatment were also investigated.

Patients with self-perceived sleep problems were offered a six-session group treatment based on CBT-i. The primary outcome was clinical feasibility, defined as: the influx of patients sufficient to start at least one group per semester (at least 8 patients); at least half of included patients participate in the first session; patients participate in at least half of the sessions; less than half of the patients drop out of treatment; group leaders find the treatment manual credible, easy to use and want to continue working with it after the study is completed.

Secondary outcomes were changes in insomnia symptoms, and changes in symptoms of depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient at a specialist outpatient clinic treating these patient groups
* Insomnia disorder or sleep problems of insomnia type
* Over 10 points on the Insomnia Severity Index (ISI)
* Adequate skills in written and spoken Swedish
* No practical barriers to participate in the group treatment

Exclusion Criteria:

* night shift work
* ongoing alcohol or drug abuse that required treatment at a specialised unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants registering to participate in the treatment | Screening
  Influx of patients should be sufficient to start at least one group per semester (at least 8 patients)
Number of included participants attending the first treatment session | First session (1 week)
  At least half of included patients should attend the first treatment session
Number sessions attended by the participants | Post-treatment (6 weeks)
  Average number of sessions attended should be no less than 3
Number of participants dropping out of treatment | Post-treatment (6 weeks)
  Less than half of the patients should drop out of treatment
Qualitative measure of group leaders' perception of the manual | Post-treatment (6 weeks)
  Group leaders should find the treatment manual credible and easy to use, and be willing to continue using the treatment manual after the study is completed

SECONDARY OUTCOMES:
Insomnia Severity Index | Post-treatment (6 weeks), Three-month follow-up (21 weeks)
  7-item self-reported measure of insomnia severity, 0-28 points, lower is better.
Patient health questionnaire (PHQ-9) | Post-treatment (6 weeks), Three-month follow-up (21 weeks)
  9-item depression inventory, 0-27 points, lower is better
Generalized Anxiety Disorder Assessment (GAD-7) | Post-treatment (6 weeks), Three-month follow-up (21 weeks)
  7-item anxiety inventory, 0-21 points, lower is better

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Jernelöv, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Program for Anxiety and Affective disorders, Stockholm Southwest Psychiatry, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cassel M, Blom K, Gatzacis J, Renblad P, Kaldo V, Jernelov S. Clinical feasibility of cognitive behavioural therapy for insomnia in a real-world mixed sample at a specialized psychiatric outpatient clinic. BMC Psychiatry. 2022 Sep 9;22(1):600. doi: 10.1186/s12888-022-04231-4. PMID 36085009